CLINICAL TRIAL: NCT00907023
Title: The Transition From Hospital to Home in Parents of Solid Organ Transplant Recipients
Brief Title: Transition From Hospital to Home in Solid Organ Transplant (SOT)
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Stacee Lerret, RN, CPNP, Medical College of Wisconsin
Other Study IDs: CHW 09/10; GC 811
Record Dates: First submitted 2009-05-20; First posted 2009-05-22 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Solid Organ Transplant
Keywords: solid organ transplant; hospital discharge

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SOT: Patients that have had a solid organ transplant

SUMMARY:
The aim of this study is to determine the influences of discharge teaching and care coordination on how ready a parent is to take their child home from the hospital after a solid organ (kidney, heart and liver) transplant. This study will also look into how the parent handles coping, utilization of healthcare resources, and parent adjustment 3 weeks after discharge from the hospital.

DETAILED DESCRIPTION:
Parents of children that have received a heart, kidney or liver transplant will be asked to participate in this protocol. Involvement in this study involves completion of questionnaires prior to the child being discharged from the hospital. Three weeks after discharge, there will also be a follow-up phone call to complete more questionnaires.

Readiness for hospital discharge is a under-investigated topic in pediatric solid organ transplant patients, despite the increasing number of pediatric patients undergoing transplant surgery. Results from this study will be used to develop an intervention program to promote readiness for hospital discharge in parents of children who receive a solid organ transplant.

ELIGIBILITY:
Inclusion Criteria:

* parents of children who have undergo a heart, kidney, or liver transplant
* English Speaking
* Parents are 18 years of age or older

Exclusion Criteria:

* parents with significant cognitive or communication impairment that would not allow them to complete the questionnaires
* parent whose child is receiving their 2nd or 3rd organ transplant

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Three Pediatric Transplant Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2009-01; Primary Completion 2010-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Determine the influences of care coordination and discharge teaching on readiness for discharge in solid organ transplant recipients | 2 years

SECONDARY OUTCOMES:
Determine the relationship of parent readiness for hospital discharge with coping, utilization of healthcare resources, medication adherence, and parent adjustment following hospital discharge | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Stacee Lerret, CPNP, Principal Investigator — Medical College of Wisconsin
Locations (3):
- United States (3):
  - Children's Memorial Hospital, Chicago, Illinois
  - Levine Children's Hospital, Charlotte, North Carolina
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin